CLINICAL TRIAL: NCT02195622
Title: Randomized Controlled Trial Comparing Two Different Morcellators for HoLEP Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana Kidney Stone Institute (Other)
Collaborators: Richard Wolf Medical Instruments Corporation (RWMIC) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1305011478R001
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Benign Prostatic Hypertrophy Requiring Surgical Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lumenis VersaCut Morcellator (Other): Lumenis VersaCut Morcellator will be utilized for prostate tissue morcellation
  Interventions: Device: Lumenis VersaCut Morcellator
- Wolf Piranha Morcellator (Other): Wolf Piranha Morcellator will be utilized for prostate tissue morcellation
  Interventions: Device: Wolf Piranha Morcellator

INTERVENTIONS:
Device: Lumenis VersaCut Morcellator
  Arms: Lumenis VersaCut Morcellator
Device: Wolf Piranha Morcellator
  Arms: Wolf Piranha Morcellator

SUMMARY:
To compare efficiency, in terms of tissue morcellation and removal time, of two commercially available FDA-approved morcellators: the VersaCut and the Piranha in subjects undergoing HoLEP procedure for benign prostatic hyperplasia (BPH).

DETAILED DESCRIPTION:
Holmium laser enucleation of the prostate (HoLEP) with mechanical morcellation is a surgical technique used for treatment of bladder outlet obstruction (BOO) secondary to benign prostatic hyperplasia (BPH). HoLEP represents a state of the art alternative to transurethral resection of the prostate (TURP). HoLEP has been shown to be safe and effective for treating prostates of all sizes and has low perioperative morbidity.

A holmium laser fiber is passed through a continuous-flow resectoscope and is used to resect the obstructing prostate tissue (enucleation). After enucleation is performed, the resected tissue is advanced into the bladder. The morcellator is then used to cut the tissue into small pieces which are then removed from the bladder via suction through the morcellator blades (morcellation). We currently use the first commercially available morcellator (VersaCut, Lumenis Incorporated, Santa Clara, CA). The Storz continuous-flow resectoscope (Karl Storz,Tuttlingen, Germany) is currently used to perform the enucleation portion of the procedure.

Recently, a new morcellator has been developed (Piranha, Richard Wolf, Knittlingen, Germany). The Wolf morcellator has been reported to remove tissue at a faster rate than the Lumenis device

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo HoLEP for bladder outlet obstruction due to the prostate.
* Able to give informed consent.
* Age 18 years or older

Exclusion Criteria:

* • Inability to give informed consent.

  * Age less than 18 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-09; Primary Completion 2015-01 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- IU Health Physicians Urology, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lumenis VersaCut Morcellator: Lumenis VersaCut Morcellator will be utilized for prostate tissue morcellation
  Lumenis VersaCut Morcellator
- Wolf Piranha Morcellator: Wolf Piranha Morcellator will be utilized for prostate tissue morcellation
  Wolf Piranha Morcellator
Period: Overall Study
Arm/Group | Lumenis VersaCut Morcellator | Wolf Piranha Morcellator
Started | 37 | 37
Completed | 37 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lumenis VersaCut Morcellator | Wolf Piranha Morcellator | Total
Number analyzed (Participants) | 37 | 37 | 74
Age, Continuous [Mean (Full Range); unit: years] | 68 [45 to 88] | 69 [50 to 84] | 68.5 [45 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 37 | 37 | 74
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 37 | 37 | 74

OUTCOME MEASURES:

1. Primary Outcome: Morcellation Rate
Description: Operatively, the amount of enucleated tissue removed (in grams) per the time for complete removal (in minutes) will be recorded as "morcellation rate."
Time Frame: Collected intraoperatively upon completion of enucleation (surgical removal) of the extra benign prostate tissue growth
Measure: Mean (Full Range); unit: grams/minute
Arm/Group | Lumenis VersaCut Morcellator | Wolf Piranha Morcellator
Number analyzed (Participants) | 37 | 37
grams/minute | 4.8 [1.3 to 9.5] | 5.6 [1.4 to 18]

ADVERSE EVENTS:
Time Frame: adverse event data collected intraoperatively through hospital discharge, which is typically less than 24 hours total
Arm/Group | Wolf Piranha Morcellator | Lumenis VersaCut Morcellator
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No